CLINICAL TRIAL: NCT05114304
Title: Prevalence of Mood and Anxiety Disorders in Adult Patients With Pulmonary Langerhans Cell Histiocytosis: an Exploratory Study
Brief Title: Prevalence of Mood and Anxiety Disorders in Adult Patients With Pulmonary Langerhans Cell Histiocytosis
Acronym: PsyHistio
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210292
Record Dates: First submitted 2021-10-18; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Langerhans Cell Histiocytosis
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Langerhans cell histiocytosis (PLCH): Adults with pulmonary Langerhans cell histiocytosis
  Interventions: Other: Evaluation of co-morbid psychiatric disorders

INTERVENTIONS:
Other: Evaluation of co-morbid psychiatric disorders — Added scales :
  * Mini Internationnal Neuropsychiatric Interview
  * Fagerström test
  * DSM-5 Scale
  Additional dosage : - a urine sample will be taken to evaluate the presence of tobacco and nicotine breakdown products and the presence of various toxics
  Expired carbon monoxide for patients using nicotine substitutes

SUMMARY:
Pulmonary Langerhans cell histiocytosis (PLCH) is a rare disease, of unknown etiology, that occurs almost exclusively in smokers.The clinical experience suggests a high prevalence of anxiety symptoms and an addictive profile. However, no study to date has precisely investigated the prevalence of co-morbid psychiatric disorders in this population.The aim of the study is to evaluate the prevalence of co-morbid psychiatric disorders in adult PLCH patients.

This study should allow:

* to assess the prevalence of psychiatric disorders co-morbid in PLCH patients
* a targeted and more effective management of patients
* a better response rate to smoking and cannabis weaning, that represents a major goal for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years of age or older with PLCH diagnosed at adulthood
* Patients affiliated to the French Health Care System
* Informed patients

Exclusion Criteria:

* Patient unable to understand the interview (language barrier)
* Patient under guardianship or curatorship
* Patient under AME (French medical help for foreigners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with pulmonary Langerhans cell histiocytosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with at least one of the disorders detailed in the Mini International Neuropsychiatric Interview (MINI) test | at inclusion
  The Mini-International Neuropsychiatric Interview (M.I.N.I.) is a structured diagnostic interview (40 minutes duration), exploring in a standardized way the main psychiatric disorders of Axis I of the DSM-IV TR (American Psychiatric Association), namely 14 items with a binary result for each specified disorder

SECONDARY OUTCOMES:
Proportion of patients with at least one comorbid addictive disorder among: tobacco, alcohol, cannabis, benzodiazepines, cocaine, opiates | at inclusion
  Definition and diagnosis of addictive disorder will be assessed with Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5)
Proportion of patients with active tobacco consumption with or without comorbid psychiatric disorder | at inclusion
  Tobacco consumption will be assessed by Fagerström survey and DSM-5, cotinine in urine quantification and expired carbon monoxide for patients using nicotine substitutes. Fargerstrom test evaluates the dependence on cigarettes from 0 to 10 (0 indicated a very low dependence and 10 a very strong dependence)
Proportion of patients with persistent tobacco consumption despite nicotine replacement treatment | at inclusion
  Tobacco consumption will be assessed by Fagerström survey and DSM-5 and expired carbon monoxide for patients with nicotine substitutes
Number of previous tobacco weaning episodes and co-morbid psychiatric disorders | at inclusion
Number of co-morbid psychiatric disorders | at inclusion
Factors associated with psychiatric disorders as assessed by Mini International Neuropsychiatric Interview (MINI) test | at inclusion
  The Mini-International Neuropsychiatric Interview (M.I.N.I.) is a structured diagnostic interview (40 minutes duration), exploring in a standardized way the main psychiatric disorders of Axis I of the DSM-IV TR (American Psychiatric Association), namely 14 items with a binary result for each specified disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint-Louis, Centre de référence national des histiocytoses, Service de Pneumologie, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided